CLINICAL TRIAL: NCT01677676
Title: A Randomised, Double-Blind, Double Observer, Study to Assess the Safety, Tolerability and Immunogenicity of Repeated Intramuscular Administration of Two Different Formulations of an Influenza A Vaccine (FP-01.1)
Brief Title: Safety, Tolerability and Immunogenicity of Two Different Formulations of an Influenza A Vaccine (FP-01.1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immune Targeting Systems Ltd (Industry)
Collaborators: INCResearch Australia Pty Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FP-01.1_CS_02
Record Dates: First submitted 2012-08-24; First posted 2012-09-03 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Influenza A
Keywords: Influenza A
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 2 (Active Comparator): FP-01.1 (250µg/peptide)
  Interventions: Biological: FP-01.1
- Group 3 (Active Comparator): FP-01.1-Adjuvant (150µg/peptide / 10.8mg)
  Interventions: Biological: FP-01.1-Adjuvant
- Group 4 (Active Comparator): FP-01.1-Adjuvant (250µg/peptide / 18mg)
  Interventions: Biological: FP-01.1-Adjuvant
- Group 1 (Active Comparator): FP-01.1 (150µg/peptide)
  Interventions: Biological: FP-01.1

INTERVENTIONS:
Biological: FP-01.1 — IM injection
  Other Names: Flunisyn
  Arms: Group 1; Group 2
Biological: FP-01.1-Adjuvant — IM injection
  Other Names: Flunisyn + Adjuvant
  Arms: Group 3; Group 4

SUMMARY:
This study has been designed to evaluate the safety and immunogenicity of two different formulations of FP-01.1 as well as build on the data set from the first in human study FP-01.1_CS_01. It is anticipated that the results of this Phase I study will inform the best formulation of the vaccine to evaluate in efficacy studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 55 years inclusive at the time of consent
2. Willing to comply with the applicable contraceptive requirements of the protocol

   • For male subjects, agreement to use a barrier method (condom) as a method of birth control in addition to any contraceptive measures normally taken by his partner until completion of the Day 57 visit, and refrain from fathering a child at least until completion ofthe Day 57 visit. Male subjects do not need to use contraception if their partner has been through the menopause, or has had her womb or both her ovaries removed.

   OR

   • For female subjects of childbearing potential, be surgically sterile or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the TGA combined with a barrier contraceptive through to completion of the Day 57 visit study and have negative results on a serum or urine pregnancy test done before administration of study medication (women who are postmenopausal [no menses for at least 2 years] are also eligible to participate)
3. Satisfactory medical assessment with no clinically significant or relevant abnormalities in medical history, physical examination, vital signs, ECG and laboratory evaluation (haematology, biochemistry or urinalysis) as assessed by the Investigator.
4. An understanding, ability and willingness to fully comply with study procedures and restrictions
5. Ability to provide written, personally signed and dated informed consent to participate in the study.
6. The subject has a body mass index (BMI) within the range 19.0-32.0 kg/m2 and falls within the weight range of 50.0-100.0 kg.
7. The subject is willing to present a study prepared letter to a General Practitioner (GP) if visiting for any purpose
8. Subject is willing to refrain from consuming alcohol for 24h prior to all visits.

Exclusion Criteria:

1. As a result of the medical screening process, the Principal Investigator or Co-Investigator considers the subject unfit for the study.
2. Current, chronic or recurrent disease (e.g. cardiovascular, respiratory, endocrine, renal, liver, gastrointestinal, autoimmune, immune suppression, malignancy or other conditions) that could affect the action, absorption or disposition of the IMP or could affect clinical or laboratory assessments.
3. Significant illness as judged by the Principal Investigator or Co-Investigator within 2 weeks of the first dose of IMP.
4. Subjects with a history of allergies or allergic conditions including anaphylactic reactions, asthmatics, hay fever and eczema sufferers requiring medication which in the opinion of the Principal Investigator or Co-Investigator will affect their participation in the study.
5. Subjects receiving medications that affect the immune system including systemic steroids and patients on chronic medications where the dose has not been stable for at least 3 months.
6. Known or suspected intolerance or hypersensitivity to the IMP, or closely related compounds or any of the stated ingredients
7. History of alcohol or other substance abuse within the last year. A positive screen for alcohol or drugs of abuse.
8. Male subjects who consume more than 21 units of alcohol per week and female subjects who consume more than 14 units of alcohol per week.
9. A positive HIV antibody screen, Hepatitis B surface antigen, Hepatitis B core antibody, or Hepatitis C antibody screen
10. Subjects who have significant scarring, tattoos, abrasions, cuts or infections, that in the opinion of the Investigator could interfere with evaluation of injection site local reactions, over the deltoid region of both arms as these will be the dose site.
11. Donation of blood or blood products (e.g. plasma, platelets) within 90 days prior to or intention to donate blood during the entire study.
12. Use of another investigational medicinal product within 90 days prior to receiving the first dose of IMP or intention to enrol in another clinical study throughout the entire study (up to and including Day 57), including the 6 month follow-up period for those subjects who consent to remain on study for this follow-up.
13. Subject with suspected recent (≤12 months) pre-exposure to the influenza A virus - flu like symptoms associated with ≥ 2 days off normal daily activities
14. Subjects who have received a flu vaccine in the last 12 months or who anticipate receiving it within the duration of the clinical phase of the study (ie up to completion of Day 57) or the period up to the 6 month safety follow-up telephone call, for the subjects who consent to remain on study for this follow-up.
15. Any clinically significant abnormalities, in the opinion of the Principal Investigator or Co-Investigator, on electrocardiograms (ECGs), as assessed against the clinical site's reference range.

In addition, for each subject, a completed medical history questionnaire will be taken as part of the consented study procedure.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number and proportion of subjects reporting solicited local reactions and severity of the local reactions | Day 1-57
To assess and compare the immunogenicity response between groups | Day 1-57
  The immunogenicity of two different formulations of FP-01.1 after each vaccine injection in each treated group
Number and proportion of subjects reporting solicited systemic events | Day 1-57, optional safety FU day 209
Number and proportion of subjects reporting unsolicited AEs and Serious Adverse Events (SAEs) | Day 1-57, optional safety follow up at day 209
Number and proportion of subjects with abnormal haematology, blood chemistry lab assessments | Day 1-57
Number and proportion of subjects with abnormal vital signs/ECG assessments | Day 1-57

SECONDARY OUTCOMES:
Exploratory immunogenicity tests on samples obtained from subjects | Day 1-57
  Additional assessment of T cell responses induced by the vaccine including virus strain cross reactivity and intracellular cytokine staining assays.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Marjason, Principal Investigator — Q-Pharm Pty Ltd
Locations (1):
- Q-Pharm Pty Ltd, Brisbane, Queensland, Australia